CLINICAL TRIAL: NCT00384722
Title: EASYTRAK® 3 Downsize Lead Clinical Investigation
Brief Title: EASYTRAK 3 Downsize Lead
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Steven McQuillan, Director of Clinical Affairs, Boston Scientific
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Clinicals0011
Record Dates: First submitted 2006-10-03; First posted 2006-10-06 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2009-06

CONDITIONS: Heart Failure
Keywords: Left ventricular lead; Pacing; Heart Failure
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Device: EASYTRAK 3 Downsize Lead — EASYTRAK 3 Downsize Lead

SUMMARY:
The primary objective of this clinical investigation is to evaluate the safety and effectiveness of the EASYTRAK 3 Downsize Lead.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, multi-center US clinical investigation, designed to demonstrate the safety and effectiveness of the Guidant EASYTRAK 3 Downsize Lead in humans.

ELIGIBILITY:
Inclusion Criteria:

* Must be indicated for a Guidant CRT-P or CRT-D device
* Creatinine < 2.5 mg/dL obtained no more than two weeks prior to enrollment
* Age 18 or above, or of legal age to give informed consent specific to state and national law
* Willing and capable of providing informed consent, undergoing a device implant, participating in all testing associated with this clinical investigation at an approved clinical investigation center and at the intervals defined by this protocol
* Geographically stable residents who are available for follow-up

Exclusion Criteria:

* Have a known hypersensitivity to a 0.5 mg nominal dose of dexamethasone acetate
* Have or had previous cardiac resynchronization therapy, a coronary venous pace/sense lead or attempted LV lead placement
* Have pre-existing cardioversion/defibrillation leads or right ventricular pacing leads other than those specified in the investigational plan (unless the investigator intends to replace them with permitted cardioversion/defibrillation leads)
* Currently requiring dialysis
* Have had a myocardial infarct, unstable angina, percutaneous coronary intervention, or coronary artery bypass graft during the preceding 30 days prior to enrollment
* Have hypertrophic obstructive cardiomyopathy or infiltrative cardiomyopathy (e.g., amyloidosis, sarcoidosis)
* Documented life expectancy of less than six months or expected to undergo heart transplant within the next six months
* Enrolled or participating in any concurrent study, including drug investigations, without Guidant written approval, that may confound the results of this study
* Have a pre-existing unipolar pacemaker that will not be explanted/abandoned
* Have a mechanical tricuspid heart valve
* Women who are pregnant or plan to become pregnant. Note: Women of childbearing potential must have a negative pregnancy test within seven days of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-03; Primary Completion 2006-07 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Lead-related complication-free rate at one-month | 1 month
Chronic mean pacing thresholds at one-month. | 1 month

SECONDARY OUTCOMES:
Chronic mean R-wave amplitudes at one-month | 1 month
Chronic mean pacing impedances at one-month. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: John Hummel, MD, Principal Investigator — Riverside Methodist Hospital
Locations (1):
- Multiple Locations, Saint Paul, Minnesota, United States

REFERENCES:
- See also: Heart Failure — http://www.nlm.nih.gov/medlineplus/